CLINICAL TRIAL: NCT01254825
Title: The Efficacy of Adductor-Canal-Block (ACB) in Patients After Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Malene Espelund, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-ME-10
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Meniscus Lesion; Pain (Knee); Diagnostic Knee Artroscopy; Minor Knee Surgery
Keywords: Adductor Canal Block (ACB); Diagnostic Knee Arthroscopy; Saphenous nerve; Pain; Ultrasound block
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor-Canal-Block, Ropivacain (Experimental): Adductor-Canal-Block, 30 mL Ropivacain 7,5 mg/mL. Single dose. Ultrasound-guided application. 36 patients
  Interventions: Procedure: Adductor-Canal-Block, Ropivacain
- Adductor-Canal-Block (ACB) - Saline (Placebo Comparator): Adductor-Canal-Block, Placebo (30 mL Saline). Ultrasound-guided application. 36 patients.
  Interventions: Procedure: Adductor Canal Block, Placebo (saline)

INTERVENTIONS:
Procedure: Adductor-Canal-Block, Ropivacain — Ultrasound-guided ACB; 30 mL Ropivacain 7,5 mg/mL. Single dose.
  Other Names: Naropin (Ropivacain)
  Arms: Adductor-Canal-Block, Ropivacain
Procedure: Adductor Canal Block, Placebo (saline) — Ultrasound-guided Adductor Canal Block; 30 mL Saline. Single dose.
  Arms: Adductor-Canal-Block (ACB) - Saline

SUMMARY:
The Purpose of this study is to determine whether Adductor-Canal-Block (ACB) is superior to placebo when it comes to analgetic efficacy after Knee-Arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Knee-arthroscopy
* Written consent
* ASA I-III
* BMI 19-35

Exclusion Criteria:

* Unable to communicate in Danish
* Allergic reactions toward drugs used in the trial
* Pregnancy
* Abuse of alcohol/drugs
* Daily opioid intake
* Infection at injection site
* Can not be mobilised to 5 meters of walk; pre-surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain-Score (VAS) - patient standing | 2 hours postoperative
  Pain-score messured on a Visual Analog Scale (VAS) 2 hours after adductor canal block. Patient standing. Intervention-group vs. placebo-group.

SECONDARY OUTCOMES:
Pain-score (VAS), patient at rest | 0,1,2,4,6,8,24 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient standing | 1,2,4,6,8,24 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), after 5 meters of walk | 2,4,6,8,24 hours postoperative
  ACB-group vs. placebo
Total Opioid-consumption | 0-24 hours postoperative
  ACB-group vs. placebo-group
Opioid-consumption, postoperative | 0-2, 2-4, 4-6, 6-8, 8-24 hours postoperative
  i.v. morfin 0-2 hours postoperative tbl. morfin 2-24 hours postoperative ACB vs. placebo
Postoperative Nausea and vomiting | 0-1, 1-2, 2-4, 4-6, 6-8, 8-24 hours postoperative
  Rating-scale 0-3 ACB-group vs. placebo-group
Postoperative ondansetron consumption | In-hospital
  ACB-group vs. placebo-group
Sedation | 0,1,2,4,6,8,24 hours postoperative
  Rating-scale: 0-3 ACB-group vs. placebo-group

CONTACTS AND LOCATIONS:
Overall Officials: Malene Espelund, MD, Principal Investigator — Glostrup University Hospital, Copenhagen, Denmark
Locations (1):
- Department of Anaesthesiology, Glostrup University Hospital, Glostrup Municipality, Copenhagen, Denmark

REFERENCES:
- [Derived] Espelund M, Fomsgaard JS, Haraszuk J, Dahl JB, Mathiesen O. The efficacy of adductor canal blockade after minor arthroscopic knee surgery--a randomised controlled trial. Acta Anaesthesiol Scand. 2014 Mar;58(3):273-80. doi: 10.1111/aas.12224. Epub 2013 Nov 8. PMID 24205802